CLINICAL TRIAL: NCT03117114
Title: Endocuff Vision Assisted vs. Standard Polyp Resection in the Colorectum
Acronym: EVASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EVASTA
Record Dates: First submitted 2017-04-08; First posted 2017-04-17 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Colon Polyp
Keywords: colonoscopy; polyp; resection
MeSH Terms: conditions — Colonic Polyps; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Other): Standard colonoscopy without mounted Endocuff Vision device. Therefore standard polypectomy in case of polyp resection.
  Interventions: Other: Standard polypectomy
- Endocuff Vision Arm (Active Comparator): Endocuff Vision device mounted to the endoscope prior to the beginning of the procedure. Therefore EVD assisted polypectomy in case of polyp resection.
  Interventions: Device: Endocuff Vision assisted polypectomy

INTERVENTIONS:
Device: Endocuff Vision assisted polypectomy — EVD mounted to the tip of the endoscope, therefore EVD assisted polypectomy
  Arms: Endocuff Vision Arm
Other: Standard polypectomy — Absence of an EVD, standard polypectomy
  Arms: Standard Arm

SUMMARY:
Adenomas are premalignant polyps of the colon that should be resected endoscopically. Complete resection of adenomatous polyps is the major task of colonoscopy. In some cases polyp may be poorly accessible making endoscopic resection difficult. Polypectomy may be conducted using the so-called piece meal technique in these cases. However, leaving polyp residual polyps in the colon bears the risk of malignant degeneration as colorectal cancer may arise form adenomatous remnants. In case of difficult polyp locations endoscopic resection may also be time consuming. On the other hand endoscopists are facing an increased time pressure due to rising numbers of procedures during the last decades.

The Endocuff Vision device (EVD) is a cap that can be mounted to the tip of a standard endoscope. The EVD has small flexible branches on its outside. The branches turn out during withdrawal. By that the branches are getting in contact with colonic wall. This mechanism leads to a more stabilized position of the colonoscope in the bowel. It is hypothesized that resection circumstances may be improved by using an EVD. In addition, stabilizing the scope during resection may result in a reduced time effort. Until now no controlled trials exist investigating the effect of EVD on the time effect during polyp resection. Therefore a randomized controlled trial needed comparing standard polypectomy versus polypectomy using the EVD during routine colonoscopy procedures.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* age ≥ 40 years

Exclusion Criteria:

* American Society of Anesthesiologists class IV or higher
* pregnant women
* indication for colonoscopy: inflammatory bowel disease
* indication for colonoscopy: polyposis syndrome
* indication for colonoscopy: emergency colonoscopy e.g. acute bleeding
* contraindication for polyp resection e.g. patients on warfarin

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Polyp resection | up to 1 day (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 1 day)]
  Time of polyp resection will be measured using a stopwatch.

SECONDARY OUTCOMES:
Polyp detection | up to day 1
  a maximum of one day is expected for colonoscopy procedures
Cecal intubation time | up to day 1
  Time span until cecum is reached with the tip of the scope
Ileum intubation time | up to day 1
  Time span until ileum is reached
Total procedure duration | up to day 1
  Total procedure duration
Complications | up to day 1
  Bleeding, perforation and other complications
Propofol dosage | up to day 1
  Amount of propofol used for colonoscopy
Patient satisfaction | up to day 1
  Measured on a 10 point numeric scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar der TU München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Figura G, Hasenohrl M, Haller B, Poszler A, Ulrich J, Brown H, Abdelhafez M, Schmid RM, von Delius S, Klare P. Endocuff vision-assisted vs. standard polyp resection in the colorectum (the EVASTA study): a prospective randomized study. Endoscopy. 2020 Jan;52(1):45-51. doi: 10.1055/a-1018-1870. Epub 2019 Oct 15. PMID 31614373